CLINICAL TRIAL: NCT01955512
Title: Effect of Clopidogrel on Allergen Challenge in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RHMMED1063
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Arm given placebo
  Interventions: Drug: Placebo
- Clopidogrel (Experimental): Group given clopidogrel
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75mg daily for 7 days
  Arms: Clopidogrel
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
In asthma, breathing in an allergen, such as house dust mite induces inflammation in the airways. This process appears to involve an interaction between two different sorts of blood cells, platelets and white blood cells via a receptor called the P2Y12 receptor. The purpose of this study is to determine whether the drug clopidogrel which blocks the P2Y12 receptor on platelets, reduces inflammation following breathing in house dust mite in people with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of asthma
* Step one of treatment by GINA (2006) guidelines
* baseline FEV1 >80% predicted

Exclusion Criteria:

* current smoker
* ex smoker who quit <1 year prior to study and pack history >10 pack years
* current use of aspirin or other anticoagulant medication
* Diagnosis or documented history of bronchopulmonary aspergillosis or uncontrolled infections
* Any clinically significant cardiopulmonary abnormalities not related to pre-existing asthma
* Past or present tuberculosis, systemic lupus erythematosis or multiple sclerosis
* Any clinically significant neurological, renal, endocrine, gastrointestinal, hepatic or haematological abnormalities uncontrolled with standard treatment
* History of psychiatric, medical or surgical disorders that may interfere with study
* Clinical history suggestive of respiratory infection in month preceding study
* Alcohol or recreational drug abuse
* Diagnosis of immunodeficiency requiring treatment
* Treatment with immunomodulators (inhaled corticosteroids in two months or oral corticosteroids in six months prior to study)
* Ongoing allergen desensitisation therapy
* Regular use of sedatives, hypnotics, tranquillisers
* Positive hepatitis viral antigens or antibodies
* Blood donation within 3 months of the study
* Live immunisation <4 wks prior to study
* Inability to understand directions for study assessment
* Inability to be contacted in case of emergency
* Participation in another study at the same time or within a prior 3-month period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in sputum eosinophils following allergen challenge in the presence and absence of clopiodgorel | 8 days

SECONDARY OUTCOMES:
Provoking concentration of methacholine inducing 20% fall in forced expiratory volume in 1 second | 8 days
Change in sputum tissue factor concentration following allergen challenge in the presence and absence of clopidogrel | 8 days
Change in sputum tissue factor inhibitor concentration following allergen challenge in the presence and absence of clopidogrel | 8 days
Change in sputum thrombin activatable finbrinolysis inhibitor concentration following allergen challenge in the presence and absence of clopidogrel | 8 days
Change in sputum P-selectin concentration following allergen challenge in the presence and absence of clopidogrel | 8 days
Change in peripheral blood eosinophil and platelet counts following allergen challenge in the presence and absence of clopidogrel | 8 days
Change in urine fibrin degradation products and leukotriene E4 following allergen challenge in the presence and absence of clopidogrel | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Howarth, MD, Principal Investigator — Professor of Medicine; Christopher L Grainge, PhD MD, Study Director — Senior Lecturer in Medicine
Locations (1):
- University of Southampton Faculty of Medicine, Southampton, Hampshire, United Kingdom